CLINICAL TRIAL: NCT07398846
Title: A 12-Week Clinical Study to Evaluate the Efficacy of a Stannous Fluoride Toothpaste, Cetylpyridinium Chloride Mouthwash, and Battery Toothbrush Regimen in Reducing Established Dental Plaque and Gingivitis.
Brief Title: Efficacy of a Stannous Fluoride Toothpaste, Cetylpyridinium Chloride Mouthwash, and Battery Toothbrush Regimen in Reducing Established Dental Plaque and Gingivitis.
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Colgate Palmolive (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CRO-2025-05-PG-BTB-FL-BGS
Record Dates: First submitted 2026-01-27; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-01

CONDITIONS: Plaque
Keywords: gingivitis
MeSH Terms: conditions — Plaque, Amyloid; Gingivitis | interventions — Cetylpyridinium; cytidylyl-(3'-5')-cytidine; fluorophosphate; Supersmile; Toothpastes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Test 1 (Experimental): instructed to brush w/ full ribbon, 2x day / 2mins with toothpaste and battery toothbrush provided instructed to 2x day / Swish 20mL for 30 secs with mouthwash provided
  Interventions: Drug: 0.454%Stannous fluoride toothpaste; Drug: 0.075% Cetylpyridinium Chloride (CPC) and 0.28% zinc lactatmouthwashe
- Test 2 (Experimental): instructed to brush w/ full ribbon, 2x day / 2mins with toothpaste and battery toothbrush provided instructed to 2x day / Swish 10mL for 1min with mouthwash provided
  Interventions: Drug: 0.454%Stannous fluoride toothpaste; Drug: 0.022% Sodium Fluoride mouthwash
- Test 3 (Active Comparator): instructed to brush w/ full ribbon, 2x day / 2mins with toothpaste and manual toothbrush provided instructed to 2x day / Swish 10mL for 1min with mouthwash provided
  Interventions: Drug: 0.76% Sodium Monofluorophosphate (Na MFP) toothpaste; Drug: 0.022% Sodium Fluoride mouthwash

INTERVENTIONS:
Drug: 0.454%Stannous fluoride toothpaste — toothpaste
  Arms: Test 1; Test 2
Drug: 0.075% Cetylpyridinium Chloride (CPC) and 0.28% zinc lactatmouthwashe — mouthwash
  Arms: Test 1
Drug: 0.76% Sodium Monofluorophosphate (Na MFP) toothpaste — toothpaste
  Arms: Test 3
Drug: 0.022% Sodium Fluoride mouthwash — mouthwash
  Arms: Test 2; Test 3

SUMMARY:
To evaluate the efficacy of a stannous fluoride toothpaste, Cetylpyridinium Chloride Mouthwash, and Battery Toothbrush Regimen in Reducing Established Dental Plaque and Gingivitis.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent Form.
* Male and female subjects aged 18-70 years, inclusive.
* Availability for the twelve-week duration of the clinical research study.
* Good general health based on the opinion of the study investigator
* Minimum of 20 permanent natural teeth (excluding third molars).
* Initial gingivitis index of at least 1.0 as determined by the use of the Loe and Silness Gingival Index.
* Initial mean plaque index of at least 0.6 as determined by Rustogi Modification of the Navy plaque index.

Exclusion Criteria:

* Presence of orthodontic appliances;
* Presence of partial removable dentures;
* Oral pathology, chronic disease or tumor(s) of the soft or hard tissues of the oral cavity; 4. Advanced periodontal disease (purulent exudate, tooth mobility, and/or extensive loss of periodontal attachment or alveolar bone);
* Five or more carious lesions requiring immediate restorative treatment;
* Use of anticonvulsants, sedatives, tranquilizers, anti-inflammatory or daily analgesics within one month prior to the start of the study or scheduled to start such intake during the course of the study;
* Use of antibiotics any time during the one-month period prior to entry into the study;
* Ongoing use of medications known to affect the gingival tissues (i.e. calcium channel blockers, phenytoin, cyclosporine) and/or on any prescription medicines that might interfere with the study outcome;
* Participation in any other clinical study;
* Self-reported pregnancy and/or breastfeeding;
* Dental prophylaxis within the past three weeks prior to baseline examinations;
* Current allergies and/or history of allergic reactions to oral care products, personal care consumer products, or any of their ingredients;
* An existing medical condition that prohibits eating and/or drinking for periods up to 4 hours;
* Current smokers and/or a history of alcohol or drug abuse

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 135 (Estimated)
Dates: Start 2026-01-26 (Actual); Primary Completion 2026-04-20 (Estimated); Study Completion 2026-04-20 (Estimated)

PRIMARY OUTCOMES:
Loe-Silness Gingival Index | Baseline, 6-weeks, and 12-weeks
  score from 0 to 3 will be assigned by the examining dentist to all scoreable surfaces
Rustogi Modification of the Navy Plaque Index | Baseline, 6-weeks, and 12-weeks
  a red disclosing solution will be used to make plaque visible and improve scoring accuracy. Subjects will be instructed to swish approximately 10 drops of the solution in their mouth for 10-15 seconds before expectorating.

CONTACTS AND LOCATIONS:
Locations (1):
- Consumer Research Consulting, LLC, Melbourne, Florida, United States